CLINICAL TRIAL: NCT06672185
Title: A Phase 1 Study of ARC101 in Advanced Solid Tumors
Brief Title: ARC101 in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Third Arc Bio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARC101-P1-101
Record Dates: First submitted 2024-10-28; First posted 2024-11-04 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Cohorts (Experimental): ARC101 will be administered in escalating doses, with each dose escalation cohort assessing toxicity 21 days after the initial dose.
  Interventions: Drug: ARC101
- Dose Expansion Cohorts (Experimental): ARC101 will be administered at recommended phase 2 dose(s).
  Interventions: Drug: ARC101

INTERVENTIONS:
Drug: ARC101 — ARC101 will be administered according to an assigned dose schedule.

SUMMARY:
This first-in-human study will evaluate the safety, tolerability, pharmacokinetics, and antitumor activity of ARC101 in patients with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic solid tumor ovarian, testicular or other Claudin 6+ cancers
* Measurable or evaluable disease, per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate organ function

Exclusion Criteria:

* Active CNS involvement
* Malignancy diagnosis other than the disease under study within 2 years prior to the first dose of study drug.
* Presence of uncontrolled ascites
* Toxicity related to prior anticancer therapy that has not returned to Grade ≤1 or baseline levels
* Clinically significant pulmonary compromise
* Active autoimmune disease within 12 months prior to first dose of study drug.
* Female participant who is pregnant, breastfeeding, or plans to become pregnant or male participant who plans to father a child either while enrolled or within 90 days after the final administration of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Frequency and type of dose-limiting toxicities. | Day 1-Day 21 of the first treatment cycle
Occurrence and severity of adverse events, serious adverse events and laboratory values. | Day 1 to 100 days after the last dose of study drug.

SECONDARY OUTCOMES:
PK Assessment: Cmax of ARC101 | During the intervention/study therapy administration, approximately 1 year on average.
  Measurement of Maximum Observed Concentration
PK Assessment: Cmin of ARC101 | During the intervention/study therapy administration, approximately 1 year on average.
  Measurement of Minimum Observed Concentration
PK Assessment: Tmax of ARC101 | During the intervention/study therapy administration, approximately 1 year on average.
  Measurement of Time to Reach Maximum Concentration
PK Assessment: AUC of ARC101 | During the intervention/study therapy administration, approximately 1 year on average.
  Area under the plasma concentration versus time curve
Overall Response Rate | During the intervention/study therapy administration, approximately 1 year on average.
  Percentage of participants with best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1 and overall survival (OS)
Duration of Response | During the intervention/study therapy administration, approximately 1 year on average.
  Time from first objective response to disease progression per RECIST 1.1 or death to any cause
Progression-Free Survival | During the intervention/study therapy administration, approximately 1 year on average.
  PFS is defined as the time from the start of the treatment until objective disease progression per PFS is defined as the time from the start of the treatment until objective disease progression per RECIST 1.1 or death from any cause
Number of anti-drug antibody (ADA) Positive Participants | During the intervention/study therapy administration, approximately 1 year on average.
  Immunogenicity will be measured by the number of participants that are ADA positive.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (2):
  - START Midwest, Grand Rapids, Michigan
  - START San Antonio, LLC., San Antonio, Texas
- Australia (3):
  - Sunshine Coast University Private Hospital, Birtinya, Queensland
  - Cancer Research SA, Adelaide, South Australia
  - Cabrini Health Research, Malvern, Victoria
- Canada (2):
  - BC Cancer Research Centre, Vancouver, British Columbia
  - The Princess Margaret Cancer Centre, Toronto, Ontario
- Israel (3):
  - Rambam Medical Center, Haifa
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv